CLINICAL TRIAL: NCT05907239
Title: Effects of Focal Extracorporeal Shock Wave Therapy in the Treatment of Temporomandibular Disorders of Muscular Origin: a Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Effects of Focal Extracorporeal Shock Wave Therapy in the Treatment of Temporomandibular Disorders of Muscular Origin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Wu Tu Hsing, Director of Center of Acupuncture of Institute of Orthopaedics and Traumatology, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64637022.5.0000.0068
Record Dates: First submitted 2023-06-05; First posted 2023-06-18 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Temporomandibular Joint Disorders; Extracorporeal Shockwave Therapy
Keywords: Temporomandibular Joint Disorders; Extracorporeal Shockwave Therapy; Temporomandibular Joint Dysfunction Syndrome; High-Energy Shock Waves; Pain Management
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Agnosia

STUDY DESIGN:
Intervention Model Description: A double-blind randomized controlled clinical trial will be carried out with 50 patients in the control group and 50 patients in the intervention group. Patients will be prospectively selected at the Orofacial Pain Outpatient Clinic of the Division of Dentistry of HCFMUSP and will be referred to the Acupuncture Center of the Institute of Orthopedics and Traumatology of HCFMUSP. The control group will initially undergo treatment with guidelines for muscular temporomandibular disorders and treatment by shockwave therapy with a "placebo" applicator for 5 weeks, while the intervention group will undergo the same guidelines and treatment by shockwave therapy. focal point on the masticatory muscles during 5 sessions, once a week (totaling 5 weeks). Groups will be evaluated and compared in terms of improvement in pain and quality of life, in addition to follow-up after 1 month, 3 months and 6 months after the procedure.
Who Masked: Participant, Outcomes Assessor
Masking Description: One of the researchers will keep the randomization codes out of the patients' sight. Other medical researchers, separately, will apply the shockwaves and the placebo in a non-blinded manner. One researcher will assess the outcome measures, and will be blinded to the allocation of patients into groups throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Treatment group will undergo treatment with focal shock wave therapy for 5 weeks, with weekly sessions and guidance by a trained physiotherapist on habits, stretching and exercises for adequate strengthening and ergonomic guidelines to promote a better quality of life
  Interventions: Device: Focused Extracorporeal Shockwave Therapy
- Placebo (Placebo Comparator): Patients in the placebo group will undergo treatment with placebo focal shockwave therapy (using a dummy applicator) for 5 weeks and guidance by a trained physiotherapist on habits, stretching and exercises for adequate strengthening and ergonomic guidelines to promote a better quality of life
  Interventions: Device: Placebo Focused Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: Focused Extracorporeal Shockwave Therapy — We will apply 2000 focal shock wave impulses starting in each region of the affected masticatory muscles and looking for compromised muscles in the masticatory muscles such as: masseter, temporal, pterygoid (medial and lateral and digastric through a piezoelectric generator F7, G3 with a focus of 1.5cm in depth, frequency of 8Hz and intensity of 0.048mJ/mm² as long as it is tolerable to the patient (it can be reduced to a tolerable intensity of at least 0.018mJ/mm²) starting with a density of energy flow between 0.12 to 0.15 mJ/mm2, starting from an adaptation dose of 0.10 mJ/mm2 in the first 500 impulses. The non-stationary technique will be used, slowly moving the applicator. Shockwave therapy will be weekly, totaling five consecutive weeks.
  Arms: Treatment group
Device: Placebo Focused Extracorporeal Shockwave Therapy — We will apply 2000 focal shock wave impulses starting in each region of the affected masticatory muscles and looking for compromised muscles in the masticatory muscles such as: masseter, temporal, pterygoid (medial and lateral and digastric through a piezoelectric generator F7, G3 with a focus of 0cm depth, frequency of 8Hz and intensity of 0.048mJ/mm² with a fake gel pad applicator.
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the effectiveness of extracorporeal shock wave therapy (ESWT) in improving pain in patients with TMD pain after 5 weeks of treatment, 1 month and 3 months after the end of treatment. As secondary objectives, we plan to evaluate the effectiveness of focal shockwave therapy in relation to:

1. Range of motion (ROM) of the temporomandibular joint using goniometry after 5 weeks of treatment;
2. Degree of inflammation, using ultrasound evaluation in the temporomandibular joint relating to the degree of pain after focal shockwave therapy for 5 weeks;
3. Jaw movement (MM), joint noise (RA), joint pressure (PA) and disability index (DI) will be measured at each treatment session and after 5 weeks of treatment, 1 month and 3 months after the end of treatment in the affected joints;
4. Quality of life will be assessed using the "Short Form Health 36" questionnaire (SF-36) during the 5 weeks of treatment, 1 month and 3 months after the end of treatment;
5. Pain control medication will also be considered and compared before and after the proposed treatment for 5 weeks.

Safety will be assessed throughout the study by monitoring the incidence of study-related adverse events. All patients will be contacted periodically and encouraged to report any side effects.

DETAILED DESCRIPTION:
Introduction: Temporomandibular disorders (TMDs) are clinical conditions that affect the masticatory muscles, the temporomandibular joint (TMJ) and associated structures. Focal extracorporeal shock wave therapy (ESWT) can be used for the treatment of musculoskeletal disorders with good results in the literature and with the potential to treat muscular TMDs.

Objective: The aim of the study is to perform a double-blind randomized controlled clinical trial to evaluate the effects of focal shock wave therapy in the treatment of pain due to temporomandibular disorders of muscular origin in adults after 5 weeks of treatment, 1 and 3 months after the end of treatment.

Methods: A double-blind randomized controlled clinical trial will be carried out with 50 patients in the control group and 50 patients in the intervention group. Patients will be prospectively selected at the Orofacial Pain Outpatient Clinic of the Division of Dentistry, Instituto Central, Hospital das Clínicas, Faculty of Medicine, University of São Paulo (IC-HCFMUSP) and will be referred to the Acupuncture Center of the Institute of Orthopedics and Traumatology of HCFMUSP (IOT-HCFMUSP). The control group will initially undergo treatment with guidelines for muscular temporomandibular disorders and treatment by shockwave therapy with a "placebo" applicator for 5 weeks, while the intervention group will undergo the same guidelines and treatment by shockwave therapy. focal point on the masticatory muscles during 5 sessions, once a week (totaling 5 weeks). After the initial treatment period, the groups will be evaluated and compared in terms of improvement in pain and quality of life, in addition to follow-up after 1 month, 3 months and 6 months after the procedure.

Expected results: After the standardized treatment period of 1 weekly session in 5 consecutive weeks (totalizing 5 sessions), it is expected that there will be an improvement in the pain Visual Analogue Scale (VAS) and in the quality of life of patients with muscular TMDs. As there is a stimulus for differentiation of mesenchymal stem cells, neovascularization and release of angiogenic factors to occur, the effect of ESWT is expected to be lasting throughout the reassessments at 1 and 3 months.

Keywords: Temporomandibular Joint Disorders, Extracorporeal Shockwave Therapy, Temporomandibular Joint Dysfunction Syndrome, High-Energy Shock Waves, Pain Management

ELIGIBILITY:
Inclusion Criteria:

* Pain in the temporomandibular region;
* Myofascial pain diagnosed with or without limitation of mouth opening based on the Diagnostic Criteria for TMD (DC/TMD);
* Myofascial pain associated or not with joint abnormalities;
* Presence of moderate to severe pain: Visual Analogue Scale (VAS) >4;
* Duration of TMD pain (temporomandibular musculoskeletal) ≥3 months;
* Written granting of the informed consent form to participate in the study

Exclusion Criteria:

* Abnormality in blood clotting (coagulopathy) or using some type of anticoagulant;
* Primary malignant disease (tumors) in the treatment area;
* Acute infection of soft tissue or bone;
* Systemic infections;
* Epilepsy;
* Infiltration of corticosteroids at the application site in the last 6 weeks;
* Patient at high risk of some type of anesthesia or analgesia when it eventually has to be used;
* Polyarthritis;
* Polytrauma Local joint infections;
* Previous temporomandibular surgical treatments that compromise mastication;
* Treatment by physiotherapy, acupuncture before 3 months of performing the procedures
* Depression or other mental disorders;
* Clinical diagnosis of associated fibromyalgia;
* Associated systemic inflammatory rheumatic diseases;
* Widespread pain or pain elsewhere that predominates and overlaps with TMD muscle pain;
* Inability to understand the treatment protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale ("VAS") | 3 months
  Change of pain perception after application of focal shock wave therapy ranging from 0 (painless) to 10 (painful)

SECONDARY OUTCOMES:
Pressure pain threshold | 3 months
  Test that uses an algometer in order to define the minimum pressure that triggers pain, at pre-established points (temporomandibular region).
Range of Motion | 3 months
  Change of range of motion (ROM) of the temporomandibular joint using ruler
Quality of life assessed by the "Short Form Health 36" questionnaire (SF-36) | 3 months
  Quality of life will be assessed by the "Short Form Health 36" questionnaire (SF-36) ranging from 0 to 100
Mandibular movement and joint noise | 3 months
  Mandibular movement (MM) and joint noise (JN) will be assessed by a trained physiotherapist. The opening pattern will be evaluated through the vertical extension of mandibular movement; maximum opening without assistance; maximum opening with assistance; "overbit". Mandibular movements will be evaluated for right and left lateral excursion, in addition to referred pain in movement. Protrusions and deviations from the midline will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Wu T Hsing, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Only Study Protocol will be shared and other details of the study (Statistical analysis plan, clinical study report) at the end of recruiting phase.

REFERENCES:
- [Background] Asquini G, Pitance L, Michelotti A, Falla D. Effectiveness of manual therapy applied to craniomandibular structures in temporomandibular disorders: A systematic review. J Oral Rehabil. 2022 Apr;49(4):442-455. doi: 10.1111/joor.13299. Epub 2022 Jan 17. PMID 34931336
- [Background] Chung J, Lobbezoo F, van Selms MKA, Chattrattrai T, Aarab G, Mitrirattanakul S. Physical, psychological and socio-demographic predictors related to patients' self-belief of their temporomandibular disorders' aetiology. J Oral Rehabil. 2021 Feb;48(2):109-123. doi: 10.1111/joor.13113. Epub 2020 Oct 26. PMID 33051894
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Lipton JA, Ship JA, Larach-Robinson D. Estimated prevalence and distribution of reported orofacial pain in the United States. J Am Dent Assoc. 1993 Oct;124(10):115-21. doi: 10.14219/jada.archive.1993.0200. No abstract available. PMID 8409001
- [Background] Skarmeta NP, Pesce MC, Saldivia J, Espinoza-Mellado P, Montini F, Sotomayor C. Changes in understanding of painful temporomandibular disorders: the history of a transformation. Quintessence Int. 2019;50(8):662-669. doi: 10.3290/j.qi.a42779. PMID 31286120
- [Background] Medlicott MS, Harris SR. A systematic review of the effectiveness of exercise, manual therapy, electrotherapy, relaxation training, and biofeedback in the management of temporomandibular disorder. Phys Ther. 2006 Jul;86(7):955-73. PMID 16813476
- [Background] Shimada A, Ishigaki S, Matsuka Y, Komiyama O, Torisu T, Oono Y, Sato H, Naganawa T, Mine A, Yamazaki Y, Okura K, Sakuma Y, Sasaki K. Effects of exercise therapy on painful temporomandibular disorders. J Oral Rehabil. 2019 May;46(5):475-481. doi: 10.1111/joor.12770. Epub 2019 Feb 19. PMID 30664815
- [Background] Arber W, Kuhnlein U. [Mutational loss of the B-specific restriction in bacteriophage fd]. Pathol Microbiol (Basel). 1967;30(6):946-52. No abstract available. German. PMID 4873409
- [Background] Vervaeke K, Verhelst PJ, Orhan K, Lund B, Benchimol D, Van der Cruyssen F, De Laat A, Jacobs R, Politis C. Correlation of MRI and arthroscopic findings with clinical outcome in temporomandibular joint disorders: a retrospective cohort study. Head Face Med. 2022 Jan 7;18(1):2. doi: 10.1186/s13005-021-00305-y. PMID 34996509
- [Background] Li W, Wu J. Treatment of Temporomandibular Joint Disorders by Ultrashort Wave and Extracorporeal Shock Wave: A Comparative Study. Med Sci Monit. 2020 Jun 21;26:e923461. doi: 10.12659/MSM.923461. PMID 32564051
- [Background] Jiao K, Niu LN, Wang MQ, Dai J, Yu SB, Liu XD, Wang J. Subchondral bone loss following orthodontically induced cartilage degradation in the mandibular condyles of rats. Bone. 2011 Feb;48(2):362-71. doi: 10.1016/j.bone.2010.09.010. Epub 2010 Sep 17. PMID 20850574
- [Background] Ioppolo F, Rompe JD, Furia JP, Cacchio A. Clinical application of shock wave therapy (SWT) in musculoskeletal disorders. Eur J Phys Rehabil Med. 2014 Apr;50(2):217-30. Epub 2014 Mar 26. PMID 24667365
- [Background] Imamura M, Alamino S, Hsing WT, Alfieri FM, Schmitz C, Battistella LR. Radial extracorporeal shock wave therapy for disabling pain due to severe primary knee osteoarthritis. J Rehabil Med. 2017 Jan 19;49(1):54-62. doi: 10.2340/16501977-2148. PMID 27904912
- [Background] Iuamoto LR, Imamura M, Sameshima K, Meyer A, Simis M, Battistella LR, Fregni F. Functional Changes in Cortical Activity of Patients Submitted to Knee Osteoarthritis Treatment: An Exploratory Pilot Study. Am J Phys Med Rehabil. 2022 Oct 1;101(10):920-930. doi: 10.1097/PHM.0000000000001931. Epub 2021 Nov 18. PMID 34799508
- [Background] Santamato A, Beatrice R, Micello MF, Fortunato F, Panza F, Bristogiannis C, Cleopazzo E, Macarini L, Picelli A, Baricich A, Ranieri M. Power Doppler Ultrasound Findings before and after Focused Extracorporeal Shock Wave Therapy for Achilles Tendinopathy: A Pilot Study on Pain Reduction and Neovascularization Effect. Ultrasound Med Biol. 2019 May;45(5):1316-1323. doi: 10.1016/j.ultrasmedbio.2018.12.009. Epub 2019 Feb 8. PMID 30739723
- [Background] Moya D, Ramon S, Schaden W, Wang CJ, Guiloff L, Cheng JH. The Role of Extracorporeal Shockwave Treatment in Musculoskeletal Disorders. J Bone Joint Surg Am. 2018 Feb 7;100(3):251-263. doi: 10.2106/JBJS.17.00661. No abstract available. PMID 29406349
- [Background] Holfeld J, Tepekoylu C, Kozaryn R, Urbschat A, Zacharowski K, Grimm M, Paulus P. Shockwave therapy differentially stimulates endothelial cells: implications on the control of inflammation via toll-Like receptor 3. Inflammation. 2014 Feb;37(1):65-70. doi: 10.1007/s10753-013-9712-1. PMID 23948864
- [Background] Kuo YR, Wang CT, Wang FS, Chiang YC, Wang CJ. Extracorporeal shock-wave therapy enhanced wound healing via increasing topical blood perfusion and tissue regeneration in a rat model of STZ-induced diabetes. Wound Repair Regen. 2009 Jul-Aug;17(4):522-30. doi: 10.1111/j.1524-475X.2009.00504.x. PMID 19614917
- [Background] Kim YH, Bang JI, Son HJ, Kim Y, Kim JH, Bae H, Han SJ, Yoon HJ, Kim BS. Protective effects of extracorporeal shockwave on rat chondrocytes and temporomandibular joint osteoarthritis; preclinical evaluation with in vivo99mTc-HDP SPECT and ex vivo micro-CT. Osteoarthritis Cartilage. 2019 Nov;27(11):1692-1701. doi: 10.1016/j.joca.2019.07.008. Epub 2019 Jul 16. PMID 31323297
- [Background] Mattyasovszky SG, Langendorf EK, Ritz U, Schmitz C, Schmidtmann I, Nowak TE, Wagner D, Hofmann A, Rommens PM, Drees P. Exposure to radial extracorporeal shock waves modulates viability and gene expression of human skeletal muscle cells: a controlled in vitro study. J Orthop Surg Res. 2018 Apr 6;13(1):75. doi: 10.1186/s13018-018-0779-0. PMID 29625618
- [Background] Gupta B, Ahmed N, Sidebottom AJ. Quality of life outcomes one year after replacement of the temporomandibular joint using a modified SF36 questionnaire. Br J Oral Maxillofac Surg. 2020 Apr;58(3):304-308. doi: 10.1016/j.bjoms.2019.12.003. Epub 2020 Mar 5. PMID 32147223
- [Background] Dib-Zakkour J, Flores-Fraile J, Montero-Martin J, Dib-Zakkour S, Dib-Zaitun I. Evaluation of the Effectiveness of Dry Needling in the Treatment of Myogenous Temporomandibular Joint Disorders. Medicina (Kaunas). 2022 Feb 9;58(2):256. doi: 10.3390/medicina58020256. PMID 35208580
- [Background] Schmitz C, Csaszar NB, Milz S, Schieker M, Maffulli N, Rompe JD, Furia JP. Efficacy and safety of extracorporeal shock wave therapy for orthopedic conditions: a systematic review on studies listed in the PEDro database. Br Med Bull. 2015;116(1):115-38. doi: 10.1093/bmb/ldv047. Epub 2015 Nov 18. PMID 26585999
- [Background] Rompe JD, Meurer A, Nafe B, Hofmann A, Gerdesmeyer L. Repetitive low-energy shock wave application without local anesthesia is more efficient than repetitive low-energy shock wave application with local anesthesia in the treatment of chronic plantar fasciitis. J Orthop Res. 2005 Jul;23(4):931-41. doi: 10.1016/j.orthres.2004.09.003. PMID 16023010
- [Background] Alessandri-Bonetti G, Bortolotti F, Bartolucci ML, Marini I, D'Anto V, Michelotti A. The Effects of Mandibular Advancement Device on Pressure Pain Threshold of Masticatory Muscles: A Prospective Controlled Cohort Study. J Oral Facial Pain Headache. 2016 Summer;30(3):234-40. doi: 10.11607/ofph.1500. PMID 27472526
- See also: WMA Declaration of Helsinki - Ethical principles for medical research involving human subjects. — https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- See also: Temporomandibular Syndrome - Book — https://www.ncbi.nlm.nih.gov/books/NBK551612/